CLINICAL TRIAL: NCT04781842
Title: The Effect of a Boxing Exercise Program on Turning Speed, Gait Speed, and Functional Lower Extremity Strength in People With Parkinson Disease
Brief Title: Effect of a Boxing Program on People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Husson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUSSONPT2021CLS
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: boxing; turning speed
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Pretest-posttest control group design. The intervention group is based on retrospective data provided to the investigators. The control group will be recruited from a population where a boxing program is not available.
Who Masked: Outcomes Assessor
Masking Description: Data will be deidentified prior to be provided for data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boxing Club Group (Experimental): Participation in a weekly boxing program designed for people with Parkinson Disease
  Interventions: Other: Boxing exercise program
- Control group (No Intervention): No changes to regular physical activity during the study period

INTERVENTIONS:
Other: Boxing exercise program — Participants attended an hour long class once a week for 12 weeks. Included in class was a warm up, boxing activities including weight shifting, kicking, and punching bags, strengthening activities and a cool down.
  Arms: Boxing Club Group

SUMMARY:
This study is investigating the impact of a boxing training program on people with Parkinson Disease. The investigators were provided data for the intervention group retrospectively by the organizers of the boxing club to assess participants' benefit from participation. The outcome measures were selected to measure different aspects of functional mobility. Of particular interest is the impact of challenging whole-body activities designed for boxing and their impact on turning speed and gait. The second phase of the study will gather control group information from people with Parkinson Disease who have not participated in a boxing program to compare differences in pre-test and post-test data over a period of 12 weeks. The specific population and study design are currently pending global pandemic restrictions. Subject recruitment will involve people who have never had access to a program of this nature. An alternative population for recruitment may involve the same participants from the boxing club in a crossover study format since the boxing club has been suspended for over a year due to health and safety concerns during the pandemic. The control group of either situation would be instructed to carry on with their daily activities as usual without changing their physical activity. We hypothesize that the intervention group would show greater improvements in functional mobility compared to the control group.

DETAILED DESCRIPTION:
The effects of Parkinson Disease are progressive and cause limitations in functional mobility and quality of life. This is a disease that greatly impairs the motor system with key presentation of resting tremors, rigidity and bradykinesia. These impairments cause further deficiencies in gait and postural stability. Most notable is festinating gait that is exacerbated by direction changes and becomes a fall risk for patients. These physical limitations can manifest fear and avoidance behaviors in people that ultimately decrease quality of life. Activities that can improve balance, strength and coordination allow people to gain confidence in their ability to participate in their daily activities. The purpose of this study is to investigate the impact of a boxing training program on lower extremity functional strength, fall risk, gait speed, and turning speed for people with Parkinson Disease compared to a control group.

Data for the intervention group has been provided retrospectively by the organizers of the boxing club. This initial data was collected by volunteers of the club at the initial session and then at 12 weeks for purposes of progress reporting to the members. Data was de-identified prior to receipt by the investigators. The next phase of this study will involve recruitment of participants for a control group from areas that do not have established boxing programs. Pre- and post-tests will be conducted over a span of 12 weeks. Outcome measures for the future control group will be the same as the original tools provided by the boxing club. These measures will assess lower extremity functional strength, fall risk, gait speed and turning speed. Baseline data will be taken using 30-second sit to stand, Timed Up-and-Go, 180° turning speed, and gait speed. During the 12 week period, participants will be instructed to avoid changing their physical activity. At the end of 12 weeks the post-testing will be completed. Those participants in the control group will receive a gift card for participation in the study.

If pandemic concerns prevent the recruitment of new participants for a control group, an alternative approach will involve a cross-over design in which the original participants from the intervention group will serve as the control group. The boxing club will be approached to contact the twelve participants who provided intervention data. The boxing club has not been held since March, 2020 due to the pandemic restrictions. A control period for this group will be established over a twelve week period where they do not participate in any new changes to their physical activity. The same outcome measures will be collected at pre-test and twelve weeks later for post-testing.

Due to the nature of the in-person testing, extra precautions regarding Covid-19 have been implemented including a Covid-19 and Other Communicable Disease consent form outlining expectations of the participants as well as precautions by the investigators. These extra initiatives include appropriate facial masks and face shields by everyone involved at all times at the study site, physical distancing between investigators and participants with exceptions made for safety reasons, and any other procedures established by the study site.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease

Exclusion Criteria:

* Inability to walk without physical assistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Gait speed | 12 weeks
  Gait speed is recorded as the participant walks their comfortable walking speed on a level surface with a marked 4 meter path. The participant begins 1 meter before the start line and continues walking 1 meter past the 4 meter line to prevent acceleration and deceleration from affecting their speed.
30 Second Sit to Stand Test | 12 weeks
  The 30-second sit to stand test requires the participant to rise from a chair and sit back down without using their arms as many times as they can within 30 seconds. The number of completed rises is recorded. It is a measure of lower extremity functional strength.
Timed Up and Go Test | 12 weeks
  The Timed Up and Go Test involves having the participant rise from an arm chair, walk 10 feet around a marker on the floor, and return to sitting in the chair. The time of completion is recorded.
Turning speed | 12 weeks
  Involves timing the participant as they complete a 180 degree turn around a marker.

CONTACTS AND LOCATIONS:
Locations (1):
- Husson University, Bangor, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
Anticipate sharing all data at the conclusion of the study.
Supporting Information: Study Protocol
Time Frame: The data will be available within 6 months of the conclusion of the study.
Access Criteria: Unrestricted